CLINICAL TRIAL: NCT02349360
Title: Safety, Tolerability and Host Response to Lactobacillus Johnsonii
Acronym: LJ
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201400370
Record Dates: First submitted 2014-07-02; First posted 2015-01-28 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: safety; tolerability
MeSH Terms: interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): L. johnsonii N6.2 10^10 CFU in capsule form administered for 8 weeks
  Interventions: Biological: L. johnsonii N6.2
- Placebo (Placebo Comparator): Encapsulated starch placebo administered for 8 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: L. johnsonii N6.2 — L. johnsonii N6.2 10^10 CFU in capsule form administered for 8 weeks
  Other Names: Lactobacillus
  Arms: Probiotic
Biological: Placebo — Encapsulated starch placebo administered for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine the effects of the probiotic, Lactobacillus johnsonii N6.2, on safety, gastrointestinal function, wellness, fecal bacteria and blood biomarkers in healthy individuals.

DETAILED DESCRIPTION:
Healthy adult volunteers from 18-50 years of age will be recruited through the University of Florida and randomly distributed into two groups. This study is divided into 3 phases: baseline, intervention (study treatment) and washout. Participants will receive either the probiotic or placebo during the intervention phases. During the baseline phase, blood and fecal samples will be collected about 1 week before intervention initiation. On the day of a scheduled blood draw, the participant will need to arrive fasted overnight, and a light breakfast will be provided after blood draw. Starting on day 1 of the intervention phase, a second baseline blood sample will be collected and the participant will begin the study intervention (probiotic or placebo). Participants will consume 1 capsule (probiotic or placebo) daily for 8 weeks, and blood and stool samples will be collected and processed (on or around weeks 2, 4 and 8 of the intervention phase). A Fisher Scientific commode specimen collection system will be provided for stool collections. The stool collection kit may be taken home (participants will be asked to drop off the stool within 4 hours of defecation) for fecal sample collection or may use the restroom in the clinical lab at the Food Science and Human Nutrition Building in which kits will be provided for use. In the wash-out phase, participants will not consume the capsule (either the probiotic or placebo), but will provide blood and stool samples (on or around week 12). Throughout the study, participants will provide a total of 5 stool samples and 6 blood samples. Participants will be asked to complete daily and weekly questionnaires throughout all phases of the study, which will ask about quality of life (physical functioning, mental functioning, level of sleep, etc.), gastrointestinal function, and dietary intake. These assessments will be self-reported via online questionnaires. In the event that internet access is not available for a portion of the study, paper copies of the questionnaires may be provided.

ELIGIBILITY:
Inclusion Criteria:

* To participate in the study individuals must

  * be 18-50 years old.
  * be willing to complete multiple questionnaires via computer.
  * be willing to take the probiotic or placebo capsule daily for 8 weeks.
  * be willing to provide 1 stool during weeks 0, 2, 4, 8 and 12 of the study.
  * be willing to provide blood samples at weeks -1, 0, 2, 4, 8 and 12 of the study.
  * have daily access to a computer with internet access for the entire 13-wk study.
  * be willing to provide a social security number

Exclusion Criteria:

* To participate in the study individuals must NOT

  * currently take medications for constipation, diarrhea or psychological disorders (depression, anxiety, insomnia etc.).
  * have taken antibiotics within the past four weeks prior to randomization.
  * currently take probiotic supplements and do not want to discontinue a minimum of two weeks prior to the study
  * have had or are currently being treated for any diseases or illnesses such as gastrointestinal disease (gastric ulcers, Crohn's, ulcerative colitis, etc.), chronic disease like diabetes or kidney disease, immune-compromising diseases or conditions (HIV, AIDS, hepatitis, cancer, transplant patient etc.)
  * currently receive medical treatment for stress induced symptoms/disorders
  * be a current smoker

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Food Science and Human Nutrition Dept, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marcial GE, Ford AL, Haller MJ, Gezan SA, Harrison NA, Cai D, Meyer JL, Perry DJ, Atkinson MA, Wasserfall CH, Garrett T, Gonzalez CF, Brusko TM, Dahl WJ, Lorca GL. Lactobacillus johnsonii N6.2 Modulates the Host Immune Responses: A Double-Blind, Randomized Trial in Healthy Adults. Front Immunol. 2017 Jun 12;8:655. doi: 10.3389/fimmu.2017.00655. eCollection 2017. PMID 28659913
- See also: Lactobacillus johnsonii N6.2 Modulates the Host Immune Responses: A Double-Blind, Randomized Trial in Healthy Adults. — https://www.ncbi.nlm.nih.gov/pubmed/28659913

RESULTS

PARTICIPANT FLOW:
Groups:
- Probiotic: L. johnsonii N6.2 in capsule form administered for 8 weeks
  L. johnsonii N6.2: L. johnsonii N6.2 in capsule form administered for 8 weeks
Period: Overall Study
Arm/Group | Probiotic | Placebo
Started | 21 | 21
Completed | 21 | 20
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 23 [18 to 36] | 21 [18 to 48] | 21 [18 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events
Description: The number of participants reporting Adverse Events was reported.
Time Frame: 13 weeks
Population: Subjects completing the probiotic and the placebo intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Probiotic: L. johnsonii N6.2 10^10 CFU in capsule form administered for 8 weeks
  L. johnsonii N6.2: L. johnsonii N6.2 10^10 CFU in capsule form administered for 8 weeks (
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 21 | 20
Participants | 1 | 2

2. Secondary Outcome: Composite Measure of Blood Chemistry Profiles
Description: Number of clinically relevant out of range values of the comprehensive metabolic panel and hemogram during intervention through washout period vs baseline.
Time Frame: 13 weeks
Population: Subjects completing intervention and final blood draw after 4 week washout period.
Measure: Number; unit: events
Arm/Group | Probiotic | Placebo
Number analyzed (Participants) | 21 | 20
events | 0 | 0

ADVERSE EVENTS:
Arm/Group | Probiotic | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 1/21 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotic (N=21) | Placebo (N=20)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Fractured clavical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dental Abcess (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No